CLINICAL TRIAL: NCT00921752
Title: C2 -CORVUS Cholesterol-Control (C2) Controlled Targets for High Vascular Risk Patients Using Effective Statins (CORVUS)
Acronym: C2 -CORVUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-CHU-DUM-2009/1
Record Dates: First submitted 2009-06-12; First posted 2009-06-16 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Cardiovascular Risk
Keywords: Lipid therapy; high CV risk; lipid goal attainment; High cardiovascular risk patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients at high cardiovascular risk

SUMMARY:
To demonstrate a higher percent rate of achieved target lipid goals among patients at high cardiovascular risk using more potent lipid-lowering treatment options including high-potency statins and combination therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients at high cardiovascular risk according to Framingham or SCORE rates

Exclusion Criteria:

* Not eligible for lipid or statin therapy
* Intolerance to therapy
* Patients at low or intermediate CV risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory clinics
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2009-05; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Percent rate of patients achieving target LDL cholesterol goals | On each of the 3 visits performed during the study
Percent rate of patients achieving 50% or more reduction in LDL-cholesterol | On each of the 3 visits performed during the study

SECONDARY OUTCOMES:
Percent rate of patients achieving target secondary (total Ch, triglycerides, HDL Ch) goals | On each of the 3 visits performed during the study
Percent rate of compliance among patients in the study | On each of the 3 visits performed during the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Laszlo, MD, PHD, Principal Investigator — County Hospital Bekes, Gyula; Csaba Csongvai, MD, Study Director — AstraZeneca Hungary; Eva Gulyas, Study Chair — AstraZeneca Hungary
Locations (26):
- Hungary (26):
  - Research Site, Baja
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Budapest III District
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Gyöngyös
  - Research Site, Gyula
  - Research Site, Jászberény
  - Research Site, Kalocsa
  - Research Site, Karcag
  - Research Site, Kecskemét
  - Research Site, Kisvárda
  - Research Site, Mohács
  - Research Site, Nyíregyháza
  - Research Site, Orosháza
  - Research Site, Pásztó
  - Research Site, Püspökladány
  - Research Site, Salgótarján
  - Research Site, Szarvas
  - Research Site, Szekszárd
  - Research Site, Szécsény
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Tatabánya
  - Research Site, Vác

REFERENCES:
- [Background] Randomised trial of cholesterol lowering in 4444 patients with coronary heart disease: the Scandinavian Simvastatin Survival Study (4S). Lancet. 1994 Nov 19;344(8934):1383-9. PMID 7968073
- [Background] Shepherd J, Cobbe SM, Ford I, Isles CG, Lorimer AR, MacFarlane PW, McKillop JH, Packard CJ. Prevention of coronary heart disease with pravastatin in men with hypercholesterolemia. West of Scotland Coronary Prevention Study Group. N Engl J Med. 1995 Nov 16;333(20):1301-7. doi: 10.1056/NEJM199511163332001. PMID 7566020
- [Background] Sacks FM, Pfeffer MA, Moye LA, Rouleau JL, Rutherford JD, Cole TG, Brown L, Warnica JW, Arnold JM, Wun CC, Davis BR, Braunwald E. The effect of pravastatin on coronary events after myocardial infarction in patients with average cholesterol levels. Cholesterol and Recurrent Events Trial investigators. N Engl J Med. 1996 Oct 3;335(14):1001-9. doi: 10.1056/NEJM199610033351401. PMID 8801446
- [Background] Long-Term Intervention with Pravastatin in Ischaemic Disease (LIPID) Study Group. Prevention of cardiovascular events and death with pravastatin in patients with coronary heart disease and a broad range of initial cholesterol levels. N Engl J Med. 1998 Nov 5;339(19):1349-57. doi: 10.1056/NEJM199811053391902. PMID 9841303
- [Background] Downs JR, Clearfield M, Weis S, Whitney E, Shapiro DR, Beere PA, Langendorfer A, Stein EA, Kruyer W, Gotto AM Jr. Primary prevention of acute coronary events with lovastatin in men and women with average cholesterol levels: results of AFCAPS/TexCAPS. Air Force/Texas Coronary Atherosclerosis Prevention Study. JAMA. 1998 May 27;279(20):1615-22. doi: 10.1001/jama.279.20.1615. PMID 9613910
- [Background] Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol lowering with simvastatin in 20,536 high-risk individuals: a randomised placebo-controlled trial. Lancet. 2002 Jul 6;360(9326):7-22. doi: 10.1016/S0140-6736(02)09327-3. PMID 12114036
- [Background] De Backer G, Ambrosioni E, Borch-Johnsen K, Brotons C, Cifkova R, Dallongeville J, Ebrahim S, Faergeman O, Graham I, Mancia G, Manger Cats V, Orth-Gomer K, Perk J, Pyorala K, Rodicio JL, Sans S, Sansoy V, Sechtem U, Silber S, Thomsen T, Wood D; Third Joint Task Force of European and Other Societies on Cardiovascular Disease Prevention in Clinical Practice. European guidelines on cardiovascular disease prevention in clinical practice. Third Joint Task Force of European and Other Societies on Cardiovascular Disease Prevention in Clinical Practice. Eur Heart J. 2003 Sep;24(17):1601-10. doi: 10.1016/s0195-668x(03)00347-6. No abstract available. PMID 12964575